CLINICAL TRIAL: NCT06176144
Title: Impact of Desflurane Versus Sevoflurane Anesthesia Maintenance Methods on Incidence of Postoperative Delirium in Elderly Patients
Brief Title: Impact of Desflurane and Sevoflurane on Postoperative Delirium in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Min Xu, Attending anesthesiologist，Department of Anesthesiology, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Approval-No: 2023/1347
Record Dates: First submitted 2023-11-21; First posted 2023-12-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Active Comparator): Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil, sufentanil. Sevoflurane inhalation will be stopped at the end of surgery.
  Interventions: Drug: Sevoflurane
- Desflurane group (Experimental): Desflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be supplemented with remifentanil, sufentanil. Desflurane inhalation will be stopped at the end of surgery.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Desflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled desflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), and sufentanil (administered by intermittent injection).Towards the end of surgery, desflurane inhalational concentration will be decreased and sufentanil will be administered when necessary. Desflurane inhalation will be stopped at the end of surgery.
  Arms: Desflurane group
Drug: Sevoflurane — Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection).Towards the end of surgery, sevoflurane inhalational concentration will be decreased and sufentanil will be administered when necessary. Sevoflurane inhalation will be stopped at the end of surgery.
  Arms: Sevoflurane group

SUMMARY:
Advanced age is a consistent risk factor for the incidence of postoperative cognitive decline, which is associated with longer hospital stays, decreased quality of life, and increased mortality. Anaesthetic drugs can also affect postoperative cognition, as their residual effects can alter central nervous system activity. Desflurane and sevoflurane are widely used volatile anesthetics. Choice anesthetics may influence the occurrence of postoperative delirium. However, evidence in this aspect is conflicting.

DETAILED DESCRIPTION:
With increasing life expectancy, more and more patients aged 65 or older will receive general anesthesia. Rapid recovery from anesthesia may reduce the incidence of many postoperative complications, such as postoperative delirium and cognitive dysfunction. Using inhalational anesthetics is the mainstay of general anesthesia. Since they pass readily into the brain, anesthetics are usually recognized as the important cause of postoperative cognitive dysfunction. Studies have shown that inhalation anesthesia may increase the risk of postoperative delirium in elderly patients compared to propofol, but such studies mostly focus on isoflurane and sevoflurane. Concentrations isoflurane caused aggregation of amyloid peptides in cell cultures, indicating that they brought cytotoxicity to the brain; sevoflurane also showed the same cytotoxic effect. However, some studies showed that inhalational anesthetics had a protective effect on postoperative cognitive function. Desflurane is currently known to be the least biotransformation inhaled anesthetic, whose blood-gas partition coefficient is only 0.42. Desflurane is increasingly used in elderly patients in clinical practice. However, it is not clear whether general anesthesia maintained mainly by desflurane reduces postoperative delirium and early cognitive dysfunction compared with sevoflurane-based general anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years and < 90 years;
2. Scheduled to undergo non-cardiac or non-neurosurgery with an expected duration of 2 hours or more, under general anesthesia;
3. Agree to participate, and give signed written informed consent.

Exclusion Criteria:

1. Preoperative history of schizophrenia, epilepsy, parkinsonism or any diseases of central nervous system;
2. Inability to communicate in the preoperative period (coma, dementia, language barrier, impaired hearing or vision);
3. Severe diseases in cardiovascular, respiratory, liver, kidney, or preoperative American Society of Anesthesiologists physical status classification ≥ IV;
4. Alcoholism and drug dependence;
5. Other reasons that are considered unsuitable for participation by the responsible surgeons or investigators (reasons must be recorded in the case report form).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | within 7 days after surgery
  Delirium is assessed twice daily with the Confusion Assessment Method for patients without endotracheal intubation or the Confusion Assessment Method for the Intensive Care Unit for patients with endotracheal intubation.

SECONDARY OUTCOMES:
Quality of recovery, QoR15 (Quality of Recovery 15) | The day before surgery and on the 7th day after surgery or discharge
  Quality of recovery-15 questionnaire, which consists 15 questions. The score ranges from 0 to 150. The higher the score, the better the quality of recovery.
Subjective sleep quality (NRS) within 3 days after surgery. | Up to 3 days after surgery
  Subjective sleep quality is assessed once daily with the Numeric Rating Scale (an 11-point rating scale where 0 = the worst sleep and 10 = the best sleep).
Length of stay in hospital after surgery. | Up to 30 days after surgery
  Length of stay in hospital after surgery
Percentage of intensive care unit (ICU) admission after surgery. | Within 24 hours after surgery
  Percentage of intensive care unit (ICU) admission after surgery
Length of stay in ICU after surgery. | Up to 30 days after surgery
  Length of stay in ICU after surgery (in patients admitted to the ICU after surgery)
Incidence of complications within 30 days | Up to 30 days after surgery
  Complications are defined as newly occurred events that are harmful to patients' recovery and required therapeutic intervention
Intensity of pain within 3 days after surgery | Up to 3 days after surgery
  Intensity of pain is assessed twice daily (8-10 AM and 6-8 PM) with the Numeric Rating Scale (an 11-point rating scale where 0 = no pain and 10 = the worst pain).
Incidence of postoperative cognitive dysfunction (POCD) | The day before surgery and on the 7th day after surgery or discharge
  Postoperative changes in Neuropsychological Tests score compared with baseline preoperative Neuropsychological Test scores in both the groups.

OTHER OUTCOMES:
Cognitive function at 30 days after surgery | On the 30th day after surgery
  Cognitive function assessed with Telephone Interview for Cognitive Status-Modified (TICS-m)
TNF-α concentration | The day before surgery and 24 hours after surgery. Performed in part of enrolled patients.
  Blood specimens will be taken for measuring TNF-α, which is measured with liquid chromatography-mass spectrometry.
IL-6 concentration | The day before surgery and 24 hours after surgery. Performed in part of enrolled patients.
  Blood specimens will be taken for measuring IL-6, which is measured with fluorescence immunochromatography

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yang, MD,PhD, Principal Investigator — West China Hospital
Locations (1):
- Department of Anesthesiology, West China Hospital, Chengdu, Sichuan, China